CLINICAL TRIAL: NCT06417437
Title: New Non-invasive Brain-computer Interface: Theory, Technology and Application Demonstration - Studies on and Intervention for Depressed People Based on Non-invasive BCI and Application Verification
Brief Title: Non-invasive BCI and Application Verification for Depressed People
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: The Fourth People's Hospital of Chengdu (Other); Shanghai Jiao Tong University School of Medicine (Other); University of Electronic Science and Technology of China (Other); East China Normal University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022ZD0208505
Record Dates: First submitted 2024-04-23; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Depression; Major Depressive Disorder; Bipolar Depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Medication Group (Active Comparator): Patients with anhedonia will be using either Bupropion or Voxetine. Patients without anhedonia will be given SSRIs. Frequency and dosage will be guided by psychiatrist. Treatment will last 4 weeks.
  Interventions: Drug: SSRI
- Traditional rTMs Group (Experimental): In addition to medication using SSRIs, patients will be also treated with rTMS. The stimulated brain region has decided to be dlpfc. Treatment will last 4 weeks.
  Interventions: Drug: SSRI; Device: rTMS
- New rTMS Group (Experimental): In addition to medication using SSRIs, patients will be also treated with rTMS. The stimulated brain region has not been decided, but rbitofrontal cortex, cerebellum and others are considered. Treatment will last 4 weeks.
  Interventions: Drug: SSRI; Device: rTMS
- Neuro-Feedback Group (Experimental): In addition to medication using SSRIs, patients will be also treated with Neuro-Training. The process will be guided under fNIRS and monitored by EGG. Treatment will last 4 weeks.
  Interventions: Drug: SSRI; Behavioral: Neuro-Feedback
- Game-regulation Group (Experimental): In addition to medication using SSRIs, patients will be also treated with games that can regulate emotions. Details are not yet decided. Treatment will last 4 weeks.
  Interventions: Drug: SSRI; Behavioral: Game Regulation

INTERVENTIONS:
Drug: SSRI — Patients are not masked from the types of intervention they receive. Assessment will be done before and after each intervention. Each group is independent from other groups.
Device: rTMS — Patients will be treated targeting either the traditional brain region or new region.
  Arms: New rTMS Group; Traditional rTMs Group
Behavioral: Neuro-Feedback — Patients under 18 years old will first be considered this treatment before other methods.
  Arms: Neuro-Feedback Group
Behavioral: Game Regulation — Patients will learn how to play several games that can supposedly regulate or affect negative emotions.
  Arms: Game-regulation Group

SUMMARY:
Major Depressive Disorder (MDD) is a serious mental illness and public health problem that poses threat to both physical and mental health. According to statistics from WHO, it is estimated that more than 350 million people worldwide suffer from depression, with a prevalence rate of 2.1% in China, which is approximately 30 million people.

At present, due to the lack of neurobiological markers for screening and diagnosing depression, the identification and diagnosis of MDD are based on the judgment of professional doctors, and the treatment mostly relies on clinical symptoms.

In terms of treatment, medication remains the main stream for MDD. Although current methods have certain therapeutic effects, patients still suffer from various side effects and poor cognitive function.In current clinical practice, relying purely on symptomatic diagnosis and treatment is difficult to meet the needs of clinical practice, so there is an urgent need to search for neurobiological markers in depression and develop targeted non-invasive intervention technologies.

This study aims to combine advanced brain imaging technology, digital twin-brain models, multi-source information decoding technology, integrated detection and intervention technology. The target is to create two new types of non-invasive BCI systems that can regulate emotions. One is a intervention BCI system for MDD that is suitable for hospital settings with the purpose of precise physical stimulation, and the other one is an ecological BCI system that regulate emotions and intervene with depression which is suitable for both hospital settings and future family environments.

This study will collect a comprehensive collection of physiological and biochemical indicators from patients with depression and from healthy control groups, as well as multimodal information such as head surface electroencephalography, MRI, and eye movements under different brain states, to personalize the available BCI information of depression related brain regions, circuits, and networks. The study also tries to explore emotional-interactive games that can intervene with depression and build a game data base that is dedicated to MDD. Other goals include designing and establishing two new types of emotional regulation systems, which are precise external physical stimulation intervention and ecological intervention, constructing a BCI regulation system, and conducting application verification to evaluate the regulation effect.

DETAILED DESCRIPTION:
This study aims to establish a BCI regulation scheme and system for individuals with mdd, and to conduct validation for this application. Four more detailed contents are being designed, including 1. providing biological markers in brain regions, circuits, and networks that are probably related to MDD, 2. assessment models of the state of brain and multivariate signal mapping models, 3. virtual regulation paradigms, evaluations on the effect of the regulation , and 4. multimodal information collection and regulation software and hardware technologies.

Shanghai Mental Health Center, as the sponsor institution, tends to recruit MDD patients from daily outpatient service. The paticipants' personal information will be noted and then the patients will undergo different assessment on their level of depression, anxiety, anhedonia, manic state, cognitive status, effect and side effects of the current treatment, and their biological rhythm, sleep, quality of life, etc. Peripheral blood will be drawn for different potential biomarkers, as well as multimodal information such as EEG, eye movement, magnetic resonance imaging, magnetoencephalogram, fNIRS, and etc. Then compare the following laboratory indicators between depressed patients and healthy individuals such as differences in the concentration and gene expression of peripheral blood inflammatory factors, oxidative stress indicators, brain-derived neurotrophic factors, brain imaging, electrophysiology, blood oxygen and etc. The work above is to obtain specific neurobiological markers of MDD.

Intervention measures are as follows:

1. Traditional medication with SSRIs. MDD patients will be give different SSRIs medication and undergo a two-week treatment, after which the above assessments will be done again to evaluation the efficacy and side effects of the current treatment. For MDD patients with anhedonia, other medication can be considered such as Voxetine and Bupropion.
2. rTMS combined with traditional SSRIs medication. The current brain regions chosen for rTMS include dorsolateral pre-frontal cortex. In this part, the study tends to find out new potential brain regions suitable for physical treatment in MDD patients. The considered brain regions include orbitofrontal cortex, cerebellum and others. It uses a classic 8-shaped coils, butterfly coils, deep coils, etc., neural navigation to locate stimulation targets.
3. Treatment based on neurobiological feedback. In this kind of treatment, MDD patients are treated with neurobiological feedback and will be monitored by EGG to catch unique and specific brain waves that may considered only found in MDD patients. This treatment involves using different psychological paradigms including classic cognitive research paradigms to evaluate the outcome of neuron-training and cognitive function after treatment.

Other technologies used in this study includes:

1. Functional Magnetic Resonance Imaging. Brain images will be captures during different functional tasks such as emotional matching, Monetary Incentive Delay Task ( MID ). These images will be further analyzed to figure out the neuro-mechanism of MDD. We will be using 3T Siemens PRISMA, collecting data of rs-fMRI、DTI、T1、T2 and fMRI.
2. Electroencephalography. In this part, the investigators will be using the DSI-24 wireless dry electrode EEG system. Each subject will undergo EEG collection experiments, at least collecting EEG data in a resting state (with eyes closed and open).
3. Eye movement detection. Eye movement will be traced using Tobii Pro Spectrum.
4. Functional Near-Infrared Spectroscopy. Patients will perform different tasks under the monitoring of a portable fNIRS device called Nirsport2 wireless wearable NIRS imaging system. It consists of a 8-channel LED illuminator and 8-channel active sensor for fiberless optical detection. During the tasks, the device will provide the value and changes in the level of oxyhemoglobin and deoxygenated hemoglobin observed in the subjects.
5. Magnetoencephalogram. MEG is a completely non-invasive function detection technique, widely used in the development and research of brain function and the clinical diagnosis of brain diseases. MEG uses a sensitive magnetic sensor SQUID (Superconducting Quantum Interferometer), which is placed around the head to measure the abnormally weak magnetic field generated by neuronal activity. The detected magnetic signal data will then be analyzed and processed by a computer and superimposed on magnetic resonance imaging (MRI). Through software 3D imaging, the results can be more intuitive, making the MEG have extremely high temporal and spatial resolution.

MDD patients will be divided into different treatment gourds based on theirs condition and whether the chosen treatment would be the most suitable for them. All individuals will undergo the above assessments to establish a comprehensive, multimodal information data base, and finally after comparing the outcome before and after the treatment, the study tries to find out new and effective measures and validate their feasibility.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 12 years old, male or female, right-handed, Han ethnicity
* Meets the DSM-5 diagnostic criteria for depression, with HAMD-17 scores greater than 17 and YMRS scores less than 6;
* Primary school education or above, able to understand the research content, willing to participate in this study and sign an informed consent form

Exclusion Criteria:

* Concomitant or previous history of organic brain disease or severe traumatic brain injury, personal or family history of epilepsy;
* Severe abnormalities in heart, liver, and kidney function;
* Patients with severe physical illnesses;
* History of substance dependence or abuse (alcohol, cocaine, drugs, etc.);
* Patients with mental disorders caused by organic diseases, drug or alcohol induced mental disorders, and other mental disorders;
* Pregnancy or lactation period;
* Within six months, physical therapy such as MECT and TMS should be used;
* Implants of vegetative nerve stimulation;
* Individuals who have implanted electronic or metal instruments (such as pacemakers, defibrillators, stents, orthopedic plates, etc.) and undergo ventriculoperitoneal shunt surgery;
* Obvious visual and auditory impairment, unable to cooperate in completing neuropsychological and scale assessments.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
EEG power in alpha band between the depression patient group and healthy controls. | 2 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 2 weeks.
EEG power in beta band between the depression patient group and healthy controls. | 2 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 2 weeks.
MRI imaging of DLPFC between the depression patient group and healthy controls. | 2 weeks
  Changes in brain imaging from baseline in multimodal emotional data as assessed by MRI at 2 weeks.
HbO in fNIRS between the depression patient group and healthy controls. | 2 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 2 weeks.
Hb in fNIRS between the depression patient group and healthy controls. | 2 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 2 weeks.
EEG power in alpha band between the depression patient group and healthy controls. | 4 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 4 weeks.
EEG power in beta band between the depression patient group and healthy controls. | 4 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 4 weeks.
MRI imaging of DLPFC between the depression patient group and healthy controls. | 4 weeks
  Changes in brain imaging from baseline in multimodal emotional data as assessed by MRI at 4 weeks.
HbO in fNIRS between the depression patient group and healthy controls. | 4 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 4 weeks.
Hb in fNIRS between the depression patient group and healthy controls. | 4 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 4 weeks.
EEG power in alpha band between the depression patient group and healthy controls. | 8 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 8 weeks.
EEG power in beta band between the depression patient group and healthy controls. | 8 weeks
  Changes from baseline in multimodal emotional data as assessed by EEG at 8 weeks.
MRI imaging of DLPFC between the depression patient group and healthy controls. | 8 weeks
  Changes in brain imaging from baseline in multimodal emotional data as assessed by MRI at 8 weeks.
HbO in fNIRS between the depression patient group and healthy controls. | 8 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 8 weeks.
Hb in fNIRS between the depression patient group and healthy controls. | 8 weeks
  Changes from baseline in multimodal emotional data as assessed by fNIRS at 8 weeks.
The score of HAMD-17 in depression patient group and healthy controls. | 2 weeks
  Changes from baseline in the score of HAMD-17 at 2 weeks
The score of HAMD-17 in depression patient group and healthy controls. | 4 weeks
  Changes from baseline in depression patient group in the score of HAMD-17 at 4 weeks
The score of HAMD-17 in depression patient group and healthy controls. | 8 weeks
  Changes from baseline in depression patient group in the score of HAMD-17 at 8 weeks

SECONDARY OUTCOMES:
The change in the state of depression in depression patient groups | 2 weeks
  The state of depression in patient group measured by SDS(0-80) at 2 weeks.
The change in the state of agitation in depression patient groups | 2 weeks
  The state of depression in patient group measured by HCL-32(0-32) at 2 weeks.
The change in the state of depression in depression patient groups | 4 weeks
  The state of depression in patient group measured by SDS(0-80) at 4 weeks.
The change in the state of agitation in depression patient groups | 4 weeks
  The state of depression in patient group measured by HCL-32(0-32) at 4 weeks.
The change in the state of depression in depression patient groups | 8 weeks
  The state of depression in patient group measured by SDS(0-80) at 8 weeks.
The change in the state of agitation in depression patient groups | 8 weeks
  The state of depression in patient group measured by HCL-32(0-32) at 8 weeks.
The change in the state of anhedonia in depression patient groups | 2 weeks
  The state of depression in patient group measured by SHAPS(0-64) at 2 weeks.
The change in the state of anhedonia in depression patient groups | 4 weeks
  The state of depression in patient group measured by SHAPS(0-64) at 4 weeks.
The change in the state of anhedonia in depression patient groups | 8 weeks
  The state of depression in patient group measured by SHAPS(0-64) at 8 weeks.
The change in the state of anxiety in depression patient groups | 2 weeks
  The state of anxiety in patient group measured by different scales including GAD-7(0-56) at 2 weeks.
The change in the state of anxiety in depression patient groups | 4 weeks
  The state of anxiety in patient group measured by different scales including GAD-7(0-56) at 4 weeks.
The change in the state of anxiety in depression patient groups | 8 weeks
  The state of anxiety in patient group measured by different scales including GAD-7(0-56) at 8 weeks.
The change in the level of cognitive function in depression patient group | 2 weeks
  The level of cognitive function in patient group measured by RBANS at 2 weeks.
The change in the level of cognitive function in depression patient group | 4 weeks
  The level of cognitive function in patient group measured by RBANS at 4 weeks.
The change in the level of cognitive function in depression patient group | 8 weeks
  The level of cognitive function in patient group measured by RBANS at 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenghui Yi, chief physician, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No